CLINICAL TRIAL: NCT05187936
Title: Pre-clinical Models for Mesenchymal Stem Cell Therapy in Hemophilic Arthropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0640
Record Dates: First submitted 2021-10-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia A; Hemophilia B; Arthropathy
Keywords: mesenchymal stem cells; Healthly control
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Joint Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemophilia is a constitutional coagulation disorder responsible for a hemorrhagic phenotype in patients from an early age. Hemarthrosis is one of the most frequent complications in hemophiliacs and leads to the development of severe and early arthropathy, sometimes as early as childhood. To date, there is no curative treatment for these joint disorders and preventive treatments are insufficient to completely prevent joint degradation. Mesenchymal stem cells have been shown to be of therapeutic interest in the management of pathologies such as osteoarthritis and inflammatory arthritis through their anti-inflammatory, regenerative and anti-apoptotic effects. Hemophilic arthropathy is a separate condition at the border of these two diseases Our study aim to show pre-clinical interest of mesenchymal stem cell therapy in hemophilic arthropathy

ELIGIBILITY:
Inclusion criteria:

* Hemophilia A or B adult patient, with or without arthropathy
* Heathly control

Exclusion criteria:

* Antiinflammatory drug use
* immunosuppressive treatment or condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemophilia A or B patient, with or without arthropathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of surviva | 1 day
  Use of blood or its derivatives for in vitro studies using different types of cells (chondrocytes, mesenchymal stromal cells, synoviocytes,...). Evaluation of survival, proliferation, apoptosis, phenotype, function of cells using relevant tests including RT-qPCR, flow cytometry,ELISA and other dedicated biochemical assays.
Evaluation of proliferation | 1 day
  Use of blood or its derivatives for in vitro studies using different types of cells (chondrocytes, mesenchymal stromal cells, synoviocytes,...). Evaluation of survival, proliferation, apoptosis, phenotype, function of cells using relevant tests including RT-qPCR, flow cytometry,ELISA and other dedicated biochemical assays.
Evaluation of apoptosis, phenotype, function of cells | 1 day
  Use of blood or its derivatives for in vitro studies using different types of cells (chondrocytes, mesenchymal stromal cells, synoviocytes,...). Evaluation of survival, proliferation, apoptosis, phenotype, function of cells using relevant tests including RT-qPCR, flow cytometry,ELISA and other dedicated biochemical assays.
Evaluation of phenotype | 1 day
  Use of blood or its derivatives for in vitro studies using different types of cells (chondrocytes, mesenchymal stromal cells, synoviocytes,...). Evaluation of survival, proliferation, apoptosis, phenotype, function of cells using relevant tests including RT-qPCR, flow cytometry,ELISA and other dedicated biochemical assays.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre THERON, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC